CLINICAL TRIAL: NCT05397613
Title: Examining the Effectiveness of STAIR as an Alternative to DBT for Patients With Emotion Dysregulation and PTSD
Brief Title: STAIR for Trauma and Emotion Dysregulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sanno Zack, Clinical Professor, Stanford University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 64219
Record Dates: First submitted 2022-05-24; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Posttraumatic Stress Disorder; Borderline Personality Disorder; Emotion Regulation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Borderline Personality Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Patients will receive 12 weeks of STAIR immediately or after a delay of 12 weeks for the waitlist control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STAIR (Experimental): Participants will complete 1.5 hr group sessions once per week for 12 weeks of Skills Training in Affective and Interpersonal Regulation (STAIR). Participants will complete self-report measures pre, post, and at one month intervals.
  Interventions: Behavioral: STAIR
- Waitlist control (Experimental): First, participants will remain on the DBT waitlist for 12 weeks receiving no active intervention and will complete pre and post-measures. Then participants will complete 1.5 hr group sessions once per week for 12 weeks of Skills Training in Affective and Interpersonal Regulation (STAIR). Participants will complete self-report measures pre, post, and at one month intervals.
  Interventions: Behavioral: STAIR

INTERVENTIONS:
Behavioral: STAIR — Clinician led session that hones in on a particular deficit within these skills, including identifying and labeling emotions, managing emotions, tolerating distress, accepting feelings and increasing positive emotions, identifying trauma-based interpersonal schemas, identifying conflict between trauma-related feelings and goals, role plays surrounding issues of power and control, and role-plays related to developing flexibility in interpersonal situations involving power differentials. STAIR is a cognitive-behavioral treatment that addresses emotion regulation and interpersonal difficulties and their impact on daily living.

SUMMARY:
This study will examine the impact of Skills Training in Affective and Interpersonal Regulation (STAIR) group, using self-report measures, on Posttraumatic Stress Disorder (PTSD), emotional dysregulation, borderline personality disorder symptoms, global psychopathology, and access to quality mental health care. Aims include assessing the feasibility of STAIR, reducing patients' trauma and emotion dysregulation symptoms, examining whether STAIR may be used as an alternative to DBT for patients on the DBT, and improving patient satisfaction and clinic efficiency

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Have a DSM-5 diagnosis and/or symptoms for which DBT is an indicated treatment
* Meet DSM-5 criteria for a diagnosis of posttraumatic stress disorder (PTSD)
* Meet criteria at a subclinical level for BPD (a minimum of three symptoms)
* Must be able to make group commitments for attendance, safety, and sobriety during group

Exclusion Criteria:

* If currently receiving individual therapy that follows the DBT protocol or is an evidence-based trauma-focused therapy
* If the STAIR therapy group is determined to be clinically contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who complete the STAIR intervention | Week 12
  This number will include those who attend the 12 weeks of STAIR with no more than three missed sessions
Total score of patient treatment satisfaction ratings | Week 12
  Calculate the total score for each participant on the Client Satisfaction Questionnaire-8, and find the average of those scores. Scores are summed across items. Items 2, 4, 5, and 8 are reverse scored. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Frequency of participant attendance | Week 1 through Week 12
  Calculate the number of patients who attended each week of the STAIR treatment.
Change in emotion regulation total score from baseline to Week 12 | Baseline to Week 12
  Problems with emotion regulation will be assessed using the Difficulty in Emotion Regulation Scale. Total score ranges from 36 to 180. Higher scores indicate greater problems with emotion regulation.
Change in the severity of posttraumatic stress disorder symptom total score from baseline to Week 12 | Baseline to Week 12
  The severity of posttraumatic stress disorder symptoms is measured using the PCL-5. Items are rated using a 5-point likert scale ranging from 0 "not at all" to 4 "extremely." All 20 items are summed to obtain a total score (0 to 80), higher scores indicate higher severity of PTSD symptoms.
Change in Borderline symptom severity total score from baseline to Week 12 | Baseline and Week 12
  Using the Borderline Evaluation of Severity Scale comprising of 15 items using a likert scale rated from 5 "Almost Always" to 1 "Almost Never." There are three subscales that comprise this measure: (1) Thoughts and Emotions (2) Behaviors-Negative and (3) Behaviors-Positive. The total for each subscale is determined to score the BEST. The scores of subscales A and B are then added together and the total from subscale C is subtracted. A correction factor of 15 is added to yield the final score which can range from 12 (best) to 72 (worst).
Change in Borderline Symptom List-23 total score from baseline to Week 12 | Baseline and Week 12
  This measure assesses feelings and experiences commonly endorsed by patients with BPD. The 23-item scale utilizes a 5-point Likert scale ranging from 0 = "not at all" to 4 = "very strong." The BSL-23 is scored by summing up the scores for all of the items. Total score ranges from 0 to 92, with higher scores reflecting more severe borderline personality symptoms.
Change in current symptoms of psychopathology and psychological distress total score from baseline to Week 12 | Baseline and Week 12
  The Symptom Checklist-90-Revised is a 90-item multidimensional self-report symptom measure that assesses current symptoms of psychopathology and psychological distress. The items were scored on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). It assesses nine symptom dimensions (somatization, obsessive compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychoticism). Global measures are provided to summarize overall distress, and these include the Global Severity Index, Positive Symptom Distress Index, and Positive Symptom Total. Raw scores are calculated by dividing the sum of scores for a specific dimension by the number of items in the dimension. Global severity index is calculated by summing the scores of the nine dimensions and additional items, then dividing by the total number of responses. Total score ranges from 0 to 360. Higher scores indicate worsening of disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sanno Zack, PhD, Principal Investigator — Stanford Universtiy; Emily Livermore, PsyD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cloitre M, Koenen KC, Cohen LR, Han H. Skills training in affective and interpersonal regulation followed by exposure: a phase-based treatment for PTSD related to childhood abuse. J Consult Clin Psychol. 2002 Oct;70(5):1067-74. doi: 10.1037//0022-006x.70.5.1067. PMID 12362957